CLINICAL TRIAL: NCT05944380
Title: Periarticular Nerve Group (PENG) Block for Postoperative Rehabilitation in Total Hip Arthroplasty: a Randomized Controlled Trial
Brief Title: PENG Block for Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 496/20
Record Dates: First submitted 2023-02-19; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Hip Osteoarthritis; Hip Arthropathy; Hip Disease; Hip Pain Chronic
Keywords: periarticular nerve group block; total hip arthroplasty; pain management; multimodal analgesia; regional anesthesia
MeSH Terms: conditions — Osteoarthritis, Hip; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG with 20mL 0,5% Ropivacaine (Experimental): Patients will receive a preoperative ultrasound-guided pericapsular nerve group block with 20 mL of 0.5% ropivacaine. Using appropriate sterile precautions and procedural sedation with up to 2 mg IV midazolam, an ultrasound (Mindrey TE9) equipped with either a linear 15-6 megahertz (MHz) or a curvilinear 5-2 MHz transducer (habitus-dependent) used to identify the anterior inferior iliac spine, iliopubic eminence, and psoas muscle. After spinal anesthesia, a 22g 80 mm echogenic block needle (Stimuplex Ultra 360) is advanced lateral to medial, in the plane with the ultrasound beam, beneath the psoas tendon to the iliopubic eminence. 20 mL 0.5% ropivacaine is injected beneath the psoas tendon and above the iliopubic eminence in 5 mL increments with a periodic aspiration to prevent intravascular injection. The needle is withdrawn, and the needle entry site is wiped clean.
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution
- PENG block with 20mL 0,9% normal saline (Experimental): Patients will receive a preoperative ultrasound-guided pericapsular nerve group block with 20 mL of 0.9% normal saline. Using appropriate sterile precautions and procedural sedation with up to 2 mg IV midazolam, an ultrasound (Mindrey TE9) equipped with either a linear 15-6 megahertz (MHz) or a curvilinear 5-2 MHz transducer (habitus-dependent) used to identify the anterior inferior iliac spine, iliopubic eminence, and psoas muscle. After spinal anesthesia, a 22g 80 mm echogenic block needle (Stimuplex Ultra 360) is advanced lateral to medial, in the plane with the ultrasound beam, beneath the psoas tendon to the iliopubic eminence. 20 mL 0.9% normal saline is injected beneath the psoas tendon and above the iliopubic eminence in 5 mL increments with a periodic aspiration to prevent intravascular injection. The needle is withdrawn, and the needle entry site is wiped clean.
  Interventions: Drug: 0,9% normal saline

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — 20 mL 0.5% ropivacaine will be injected for the PENG block
  Other Names: Ropimol
  Arms: PENG with 20mL 0,5% Ropivacaine
Drug: 0,9% normal saline — 20 mL 0.9% normal saline will be injected for the PENG block
  Other Names: placebo
  Arms: PENG block with 20mL 0,9% normal saline

SUMMARY:
This randomized, double-blinded, placebo-controlled trial seeks to evaluate the efficacy of the pericapsular nerve group block on postoperative rehabilitation.

DETAILED DESCRIPTION:
The pericapsular nerve group, or PENG block, has been recently described and shows promise in providing analgesia to the hip joint. However, the effect of this block on postoperative rehabilitation is uncertain. This study compares a preoperative PENG block to a placebo before total hip arthroplasty under spinal anesthesia. The primary outcome measure is verticalization, walking distance, ability to go out of bed, active lifting of the limb, range of motion in the hip joint, bending range of motion, and abduction range of motion. The secondary measure is postoperative pain assessment during rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old undergoing unilateral total hip arthroplasty

Exclusion Criteria:

* refusal to participate
* < 18 yo
* Chronic opioid use
* localized infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
postoperative Numeric Pain Rating Scale in motion | Day 2
  Numeric Pain Rating Scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
postoperative Numeric Pain Rating Scale in motion | Day 3
  Numeric Pain Rating Scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
postoperative Numeric Pain Rating Scale in motion | Day 4
  Numeric Pain Rating Scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")

SECONDARY OUTCOMES:
total opioid consumption | 96 hours postoperatively
  milligrams of intravenous morphine equivalents
Time to first opioid | 96 hours postoperatively
  Hours to first administration of an intravenous opioid drug
postoperative Numeric Pain Rating Scale et rest | Day 1
  representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
postoperative Numeric Pain Rating Scale et rest | Day 2
  representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
postoperative Numeric Pain Rating Scale et rest | Day 3
  representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
postoperative Numeric Pain Rating Scale et rest | Day 4
  representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Functional assessment: getting out of bed without help | First day after surgery
  Binary assessment of motor function evaluated at the first day after surgical procedure
Functional assessment: active elevation of the operated limb | First day after surgery
  Binary assessment of motor function evaluated at the first day after surgical procedure
Functional assessment: independent verticalization- by the balcony | First day after surgery
  Binary assessment of motor function evaluated at the first day after surgical procedure
Functional assessment: walking by the balcony | First day after surgery
  Binary assessment of motor function evaluated at the first day after surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Domagalska, PhD, Principal Investigator — Department of Palliative Medicine, University of Medical Sciences, Poznań, Poland; Zbigniew Żaba, PhD, Study Chair — Department of Emergency Medicine Clinic
Locations (1):
- Poznan Univesity of Medical Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
The data presented in this study are available on request from the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December 2024
Access Criteria: The data presented in this study are available on request from the corresponding author.